CLINICAL TRIAL: NCT06940908
Title: Experience of Guillain Barré Syndrome in Childhood: A French Multicentric Qualitative Study
Brief Title: Living With Guillain-Barré Syndrome as Children.
Acronym: GUIREQUAL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0615
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Guillain Barré Syndrome; Guillain-Barré Syndrome (GBS)
Keywords: children; experience; qualitative study; quality of life
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- semi-structured interview: There are no intervention or comparison groups, as this is a non-interventional qualitative study. All participants will undergo a single semi-structured interview, conducted in a child-friendly and supportive setting (either in person at the hospital, or via secure video conferencing when necessary).

SUMMARY:
The goal of this qualitative observational study is to explore the lived experience and psychological aftermath of children who were affected by Guillain-Barré Syndrome (GBS) two to five years earlier. GBS is a rare and acute neurological condition, and while motor recovery is generally good in children, residual symptoms such as fatigue, pain, anxiety, or depression may persist and impact quality of life.

The main questions it aims to answer are:

How do children experience and recall their illness and recovery after GBS? What psychological or contextual factors might contribute to emotional distress or depressive symptoms in the years following the disease?

Participants will:

Be children aged 10 or older who had GBS two to five years prior. Participate in a 45-60-minute semi-structured individual interview during a routine follow-up visit.

Respond to a screening questionnaire for depressive symptoms (Children's Depression Inventory or Beck Depression Inventory Fast Screen).

Undergo a brief clinical examination to assess any remaining physical sequelae. Interviews will be audio recorded, transcribed verbatim, and pseudonymized. Thematic reflexive analysis will be performed following Braun and Clarke's methodology. Recruitment will continue until theoretical saturation is reached (approximately 25 participants expected) across two centers (Toulouse and Montpellier).

This study aims to generate new insights into pediatric psychological outcomes after GBS, in order to improve acute care and follow-up, and potentially guide future mental health support for affected children.

DETAILED DESCRIPTION:
Guillain-Barré Syndrome (GBS) is an acute inflammatory demyelinating polyneuropathy that can lead to significant functional impairment. Although pediatric patients typically experience more favorable motor recovery compared to adults, emerging clinical observations suggest that psychological and sensory sequelae-such as fatigue, neuropathic pain, paresthesia, anxiety disorders, and major depressive episodes-may persist long after the acute phase.

To date, no qualitative research has specifically examined how children experience GBS and its aftermath, particularly years after recovery. The GUIREQUAL study is designed to fill this gap by using qualitative methods to explore long-term psychosocial impacts among pediatric GBS survivors, and to develop hypotheses regarding psychological vulnerability post-recovery.

This is a bicentric, prospective qualitative study conducted in two pediatric neurology centers (Toulouse and Montpellier, France). Participants will be identified from hospital records and must meet strict inclusion criteria, including a confirmed diagnosis of GBS or its variants (AIDP, AMAN, Miller Fisher), with onset 2 to 5 years prior to study enrollment. Patients with chronic inflammatory demyelinating polyneuropathy (CIDP), central nervous system involvement (e.g., Bickerstaff encephalitis), or unrelated chronic neurological/orthopedic diseases will be excluded to reduce confounding factors.

The data collection process includes:

A semi-structured, face-to-face interview (45-60 minutes) conducted during a routine follow-up visit, allowing the child (with or without parental presence, depending on age) to recount their illness experience in a supportive setting.

A brief validated screening tool to assess current depressive symptoms (CDI or BDI-FS).

A short clinical assessment by an independent clinician to evaluate any remaining physical sequelae.

Interviews will be audio-recorded, transcribed verbatim, and pseudonymized for confidentiality. Thematic reflexive analysis will be conducted following the Braun & Clarke methodology. Transcripts will be coded iteratively, and themes will be developed inductively and refined throughout the study process, in accordance with qualitative research best practices. Data collection will continue until theoretical saturation is achieved (estimated at 25 participants), ensuring the robustness of thematic conclusions.

The research team will maintain a reflexive logbook to track methodological decisions, and triangulation will be employed across multiple researchers to enhance credibility. This approach is expected to yield a nuanced understanding of how children make sense of their illness experience and what psychosocial factors may contribute to long-term well-being or distress.

Ultimately, GUIREQUAL aims to generate new clinical hypotheses, inform psychosocial follow-up strategies, and potentially advocate for early mental health screening and support in pediatric GBS survivors.

ELIGIBILITY:
Inclusion Criteria:

* Children or adolescents aged 10 years or older at the time of the interview
* History of Guillain-Barré syndrome (GBS) diagnosed in childhood
* Time since acute episode: between 2 and 5 years
* Sufficient mastery of the French language to participate in a semi-structured interview
* Consent of the participant and, for minors, parental consent

Exclusion Criteria:

* Presence of a neurological disease other than GBS that may interfere with participation or interpretation of data
* Severe cognitive impairment preventing the child or adolescent from engaging in the interview

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be selected from the population of children and adolescents who experienced Guillain-Barré Syndrome (GBS) during childhood and received medical care at one of two university hospitals in southern France: Toulouse University Hospital and Montpellier University Hospital. Eligible participants will be aged 10 years or older at the time of the study and must be between 2 and 5 years post-acute GBS episode. The population includes individuals with sufficient command of the French language to engage in a semi-structured interview exploring the long-term psychosocial impact of GBS. Both male and female participants will be considered, provided they meet the inclusion criteria and give informed consent (or assent with parental consent for minors).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Child's psychological and emotional experience after Guillain-Barré Syndrome | From 6 months to 5 years after the acute Guillain-Barré episode
  The child's subjective experience will be assessed through a semi-structured individual interview conducted by a trained researcher. The outcome will explore psychological themes such as fear, anxiety, mood changes, body image, and coping strategies in the aftermath of Guillain-Barré Syndrome. Interviews will be recorded, transcribed verbatim, and analyzed using inductive thematic analysis. No standardized questionnaire will be used; the approach is entirely qualitative and descriptive.

SECONDARY OUTCOMES:
Child's perception of hospitalization and medical care during Guillain-Barré Syndrome | From 6 months to 5 years after the acute Guillain-Barré episode
  This outcome will assess how the child perceived their stay in hospital during the acute phase of Guillain-Barré Syndrome, including memories of medical procedures, communication with healthcare professionals, perceived support, and emotional reactions. Information will be gathered through semi-structured interviews, allowing the participant to freely express their lived experience. Thematic content analysis will be used to identify recurring patterns and significant narratives. Retrospective exploration from the onset of symptoms through hospital discharge.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University Hospital of Montpellier, Montpellier, Occitanie
  - University Hospital Toulouse, Toulouse, Occitanie

IPD SHARING:
Plan to Share IPD: No